CLINICAL TRIAL: NCT02594826
Title: Facilitating Cervical Cancer Screening Among Underserved Korean American Women
Brief Title: Cervical Cancer Screening Intervention Among Korean American Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fox Chase Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); American Cancer Society, Inc. (Other)
Responsible Party: Principal Investigator, Carolyn Fang, PhD, Principal Investigator, Fox Chase Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 09-804; NCI-2015-01176 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 09-804 (Other: Fox Chase Cancer Center); P30CA006927 (NIH); RSGT-09-011-01-CPPB (Other Grant/Funding Number: American Cancer Society)
Record Dates: First submitted 2015-10-31; First posted 2015-11-03 (Estimated); Results first posted 2016-10-13 (Estimated); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Cervical Carcinoma
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Culturally appropriate intervention (Experimental): Culturally appropriate, church-based intervention focused on cervical cancer and navigation assistance.
  Interventions: Behavioral: Culturally appropriate intervention
- General health education control (Active Comparator): General health and cancer education on nutrition, regular check-ups, tobacco use, and cancer screening.
  Interventions: Behavioral: General health education control

INTERVENTIONS:
Behavioral: Culturally appropriate intervention — Church-based educational intervention combined with navigation assistance
  Arms: Culturally appropriate intervention
Behavioral: General health education control — General health and cancer education
  Arms: General health education control

SUMMARY:
This is a randomized trial to evaluate the effects of a community-based intervention on increasing cervical cancer screening rates in underserved Korean American women. Due to the multiple factors that contribute to screening uptake, an educational program customized to Korean culture combined with navigation assistance may be effective in increasing the number of Korean American women who can access cervical cancer screening.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the efficacy of a culturally-appropriate educational intervention compared to a general cancer health education program in increasing cervical cancer screening among Korean American women.

SECONDARY OBJECTIVES:

I. To examine the effects of a culturally-appropriate intervention on women's knowledge, psychosocial beliefs about cervical cancer and screening, and barriers to screening compared to a general cancer health education program.

II. To examine the extent to which changes in knowledge, psychosocial beliefs, and barriers mediate the effects of the intervention on screening behavior.

OUTLINE: Participants are randomized to 1 of 2 arms.

ARM I (INTERVENTION CONDITION): Participants undergo a culturally appropriate, church-based intervention comprised of four components: 2-hour small group education sessions delivered at church sites by professional, bilingual community health educators (CHEs) that include culturally appropriate visual aids and print materials in Korean; navigation assistance, including language services, appointment scheduling, and transportation assistance from CHEs and church health workers (CHWs); referrals to Pap test sites; and a 6-month reminder letter for screening.

ARM II (CONTROL CONDITION): Participants undergo 2-hour general health and cancer education by bilingual CHEs, which covers nutrition, regular check-ups, tobacco use, and cancer screening. Participants also receive pre-existing written material produced by the American Cancer Society (ACS), National Institutes of Health (NIH), and Centers for Disease Control (CDC)., and are advised to seek regular preventive health services.

After completion of study, participants are followed up post-intervention and at 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Self-identified Korean ethnicity
* Possessing a functional telephone in the home or on person
* Anticipated presence in this geographic region for a period of one year

Exclusion Criteria:

* A current diagnosis of cervical cancer
* Have had a Pap test within the past 12 months
* Are currently adherent to doctor recommended screening interval

Min Age: 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 744 (Actual)
Dates: Start 2009-02; Primary Completion 2013-09 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: CAROLYN FANG, Principal Investigator — Fox Chase Cancer Center
Locations (1):
- Fox Chase Cancer Center, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Result] Fang CY, Ma GX, Handorf EA, Feng Z, Tan Y, Rhee J, Miller SM, Kim C, Koh HS. Addressing multilevel barriers to cervical cancer screening in Korean American women: A randomized trial of a community-based intervention. Cancer. 2017 May 15;123(6):1018-1026. doi: 10.1002/cncr.30391. Epub 2016 Nov 21. PMID 27869293

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Following eligibility screening and informed consent, women completed a baseline questionnaire, which included items on screening history and prior medical history. For a small number of women, responses on the baseline questionnaire were deemed to be inconsistent with study eligibility. Therefore, those women were excluded from further analysis.
Period: Overall Study
Arm/Group | Culturally Appropriate Intervention | General Health Education Control
Started | 347 | 358
Completed | 290 | 298
Not Completed | 57 | 60

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Culturally Appropriate Intervention | General Health Education Control | Total
Number analyzed (Participants) | 347 | 358 | 705
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.9 (9.5) | 53.9 (11.6) | 52.9 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 347 | 358 | 705
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 347 | 358 | 705
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 347 | 358 | 705

OUTCOME MEASURES:

1. Primary Outcome: Number of Women Who Receive a Pap Smear Test
Description: Number of women who receive a Pap smear test in each group
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | Culturally Appropriate Intervention | General Health Education Control
Number analyzed (Participants) | 290 | 298
participants | 209 | 30
Statistical Analysis 1: Comparison: General Health Education Control; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; This is the calculated p-value, which is adjusted for age, marital status, prior screening, health insurance, and having a healthcare provider; Odds Ratio (OR) = 35.8, 95% CI 2-sided [11.1 to 114.9]

2. Secondary Outcome: Knowledge About Cervical Cancer
Description: Women's knowledge was assessed using 10 items. For each item, women responded whether the statement was true ("Yes", "No", or "Don't know"). "Don't know" responses were scored as incorrect. Each item that was answered correctly was scored as '1'. Correct responses were summed across all 10 items. Therefore, women's knowledge scores could range from 0 (no correct responses) to 10 (all correct responses), where higher scores represent greater knowledge.
Time Frame: 12 months post-program
Population: Preliminary data cleaning revealed that of the 705 participants who were included in the primary analysis, 29 participants had failed to answer 1/3 or more of the items on the questionnaire. Therefore, due to extensive missing data, these participants were excluded from the analysis of the secondary outcomes.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Culturally Appropriate Intervention | General Health Education Control
Number analyzed (Participants) | 341 | 335
units on a scale | 6.6527 (0.1276) | 6.0258 (0.2116)
Statistical Analysis 1: Comparison: Culturally Appropriate Intervention vs General Health Education Control; The null hypothesis is that the two conditions would not differ in their knowledge following program participation. The study biostatistician conducted full regression models to examine change in knowledge (from pre- to post-program) within each group and across groups over time. The models controlled for relevant covariates; Test type: Superiority; p = 0.005, Regression, Linear; Controlling for: marital status, education, language spoken at home, health insurance, regular physician, language of physician, ever had Pap test

ADVERSE EVENTS:
Arm/Group | Culturally Appropriate Intervention | General Health Education Control
Serious Adverse Events (participants affected / at risk) | 0/290 | 0/298
Other Adverse Events (participants affected / at risk) | 0/290 | 0/298

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No